CLINICAL TRIAL: NCT00875992
Title: A Randomized Controlled Trial to Evaluate the Effectiveness of Angular Stable Locking System (ASLS) in Patients With Distal Tibial Fractures Treated With Expert Tibial Nails (ETN)
Brief Title: Trial to Evaluate the Effectiveness of Angular Stable Locking System (ASLS) in Patients With Distal Tibial Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Collaborators: Synthes Inc. (Industry)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASLS RCT 09
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Tibial Fractures
MeSH Terms: conditions — Tibial Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ETN with ASLS (Experimental): Angle stable locking of the Expert Tibial Nail using ASLS
  Interventions: Device: ETN with ASLS
- ETN with conventional locking (Active Comparator): Conventional locking of the Expert Tibial Nail using conventional locking bolts
  Interventions: Device: ETN locked with conventional locking bolts

INTERVENTIONS:
Device: ETN with ASLS — Angle stable locking of ETN using ASLS
  Arms: ETN with ASLS
Device: ETN locked with conventional locking bolts — Conventional surgical procedure
  Arms: ETN with conventional locking

SUMMARY:
In many cases, the existing locking bolts and screws in intramedullary nails do not provide sufficient stability. The play between screw and nail can result in loss of reduction and the instability due to the interfragmentary movement can result in malunions or nonunions. Therefore, an Angular Stable Locking System for Intramedullary Nails (ASLS) was developed to enhance axial and angular fracture stability. ASLS provides angular-stable fixation between nails and screws with resorbable sleeves used as dowels in the nail locking holes. Preliminary results of a pre-study show a trend towards reduced time to pain-free full weight bearing in patients being treated with ASLS. This hypothesis will be tested in the present randomized controlled study.

DETAILED DESCRIPTION:
The primary aim of the present study is to evaluate the effectiveness of the Angular Stable Locking System (ASLS) in patients with distal tibial fractures treated with Expert Tibial Nails (ETN). In many cases, the existing locking bolts and screws in intramedullary nails do not provide sufficient stability. The play between screw and nail can result in loss of reduction and the instability due to the interfragmentary movement can result in malunions or nonunions. Therefore, an Angular Stable Locking System for Intramedullary Nails (ASLS) was developed to enhance axial and angular fracture stability. ASLS provides angular-stable fixation between nails and screws with resorbable sleeves used as dowels in the nail locking holes. Preliminary results of a pre-study show a trend towards reduced time to pain-free full weight bearing in patients being treated with ASLS. This hypothesis will be tested in the present randomized controlled study.

ELIGIBILITY:
Inclusion Criteria:

* The patient is ≥ 18 years old
* The patient suffers from an acute distal third tibial fracture classified as:

AO 42 A1-A3, AO 42 B1-B3, AO 42 C1-C3, AO 43 A1-A3

* The fracture is fixed with an Expert Tibia Nail (ETN)
* The patient was able to walk without walking aid prior to the accident
* The patient is able to understand and read local language at elementary level
* The patient is willing and able to give written informed consent to participate in the study according to the CIP

Exclusion Criteria:

* The patient is legally incompetent
* Preexistent malunion or nonunion of the fracture under investigation
* Osteotomies
* The patient suffers from additional fractures of the lower extremities (Exception: ipsilateral fibular fracture)
* The patient suffers from a pathologic fracture
* The patient suffers from active malignancy
* The patient is pregnant, breast feeding or planning to get pregnant during the study period
* The patient suffers from a life-threatening condition
* The patient is affected by drug or alcohol abuse
* The patient has participated in any device related clinical trial affecting the lower extremities within the previous month
* The patient has participated in any drug related clinical trial affecting bone healing within the previous month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2009-06; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Time to pain free full weight bearing | 1 year

SECONDARY OUTCOMES:
Amount of partial weight bearing | Up to achievement of primary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Dankward Hoentzsch, MD, Principal Investigator — BG Unfallklinik Tübingen, 72076 Tübingen, Germany
Locations (8):
- Medizinische Universität, Innsbruck, Austria
- Germany (6):
  - Charité, Berlin
  - Medizinische Hochschule, Hanover
  - Universität des Saarlandes, Homburg/Saar
  - Friedrich-Schiller-Universität, Jena
  - Universitätsmedizin Mainz, Mainz
  - BG Unfallklinik, Tübingen
- Sykehuset i Vestfold HF, Tønsberg, Norway

REFERENCES:
- [Derived] Hontzsch D, Schaser KD, Hofmann GO, Pohlemann T, Hem ES, Rothenbach E, Krettek C, Attal R. Evaluation of the effectiveness of the angular stable locking system in patients with distal tibial fractures treated with intramedullary nailing: a multicenter randomized controlled trial. J Bone Joint Surg Am. 2014 Nov 19;96(22):1889-97. doi: 10.2106/JBJS.M.01355. PMID 25410507